CLINICAL TRIAL: NCT04443803
Title: Characterizing the Perioperative Epidemiology of SARS-CoV-2 (COVID-19) Spread for Quality Improvement of Perioperative Infection Control Program
Status: Completed | Type: Observational
Sponsor: Randy Loftus (Other)
Responsible Party: Sponsor-Investigator, Randy Loftus, MD, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202005391
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — OR PathTrac collection kits will be utilized for sampling of 48 specific locations/times throughout each case. These samples include:
  * 11 samples that have been routinely used for S. aureus including nasopharyngeal. Normally there are 13, but 2 samples are included in the subsequent environmental locations: the adjustable pressure-limiting valve and agent dial at baseline and case end.
  * 1 sample from the endotracheal tube tip at case end, as positive control.
  * 12 environmental locations at case end including anesthesia machine and each of the air vents,
  * 12 environmental locations matched after environmental cleaning, and
  * 12 environmental locations matched after Surfacide Helios UV-C cleaning. The Surfacide Helios UV-C cleaning robots will be used after all normal environmental cleaning of the room has taken place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In a case-series analysis, up to 20 patients undergoing elective or urgent/emergent surgery that are COVID-19 positive will be approached for patient consent.

OR PathTrac (RDB Bioinformatics, Omaha, NE 68154) collection kits will be utilized for sampling of 48 sampled time/locations per patient. Patient sampling locations will include the nasopharynx and oropharynx. Operating room environmental locations will include areas in the patient care arena such as the anesthesia machine. Samples of each location will be obtained before and after treatment with UV-C (Helios, Surfacide), germicidal, ultraviolet light and other infection control practices that are currently in place, such as utilization of preoperative chlorhexidine wipes, nasal iodine, improved hand hygiene, and improved vascular care.

UV-C light for environmental cleaning is not regulated by the FDA.

Samples will be processed by RT-PCR for presence of SARS-CoV-2 nucleic acid. Positive samples will be sent to Dr. Stanley Perlman's lab to assess viability. Samples will also be assessed for S. aureus as a process control. We will characterize the epidemiology of perioperative SARS-CoV-2 spread as a quality improvement initiative to improve our current perioperative infection control bundle and to serve as the platform for national dissemination of a perioperative COVID-19 defense strategy.

DETAILED DESCRIPTION:
The operating room schedule will be reviewed each day by a research assistant for COVID-19 positive patients. Additionally, the research assistant will receive a page for every emergency surgery that takes place in the OR.

OR PathTrac collection kits will be utilized for sampling of 48 specific locations/times throughout each case. These samples include:

* 11 samples that have been routinely used for S. aureus including nasopharyngeal. Normally there are 13, but 2 samples are included in the subsequent environmental locations: the adjustable pressure-limiting valve and agent dial at baseline and case end.
* 1 sample from the endotracheal tube tip at case end, as positive control.
* 12 environmental locations at case end including anesthesia machine and each of the air vents,
* 12 environmental locations matched after environmental cleaning, and
* 12 environmental locations matched after Surfacide Helios UV-C cleaning. The Surfacide Helios UV-C cleaning robots will be used after all normal environmental cleaning of the room has taken place.

A transmission event will be defined as 2 samples with detection of SARS-CoV-2 by RT-PCR, with samples obtained from 2 distinct, epidemiologically-related reservoirs within a surveillance unit. The OR PathTrac software platform will process transmission dynamics in order to continually summarize the epidemiology of SARS-CoV transmission, with results updated daily as case-pair data is continually entered into the program. This information will be continually displayed to identify the most common reservoir of origin, the most common transmission locations (vectors), and involvement of key portals of entry (stopcocks). These will become improvement targets with feedback provided via automated failure mode analysis reports. The research assistants will use the reports to continually optimize the interventions during the observational period. The incidence and epidemiology of transmission will be mapped before and after UV-C treatment and positive samples for SARS-CoV-2 examined for viability by a UIHC laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 years old) COVID-19 positive patient undergoing surgery requiring anesthesia and placement of a peripheral and/or central intravenous catheter.

Exclusion Criteria:

* <18 years old, Shellfish, iodine, chlorhexidine allergies, COVID-19 negative status, no anesthesia and/or placement of peripheral and/or central intravenous catheter required

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery at the University of Iowa
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Perioperative transmission of SARS-CoV-2 | 24 hours
  Sars-CoV-2 transmission event

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Loftus RW, Dexter F, Goodheart MJ, McDonald M, Keech J, Noiseux N, Pugely A, Sharp W, Sharafuddin M, Lawrence WT, Fisher M, McGonagill P, Shanklin J, Skeete D, Tracy C, Erickson B, Granchi T, Evans L, Schmidt E, Godding J, Brenneke R, Persons D, Herber A, Yeager M, Hadder B, Brown JR. The Effect of Improving Basic Preventive Measures in the Perioperative Arena on Staphylococcus aureus Transmission and Surgical Site Infections: A Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e201934. doi: 10.1001/jamanetworkopen.2020.1934. PMID 32219407